CLINICAL TRIAL: NCT05066191
Title: Impact of Gluten Contamination in Celiac Patients Clinically
Brief Title: Impact of Gluten Contamination in Celiac Patients Clinically Responsive and Unresponsive to the Gluten-free Diet
Acronym: GIP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Principal Investigator, Luca Elli, MD, PhD, Gastroenterologist, Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Other Study IDs: 169_2021
Record Dates: First submitted 2021-09-23; First posted 2021-10-04 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-09

CONDITIONS: Celiac Disease
Keywords: non celiac gluten sensitivity; gluten reintroduction; GIP
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — urinary and fecal samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary aim of the study is to detect the presence of gluten immunogenic peptides (GIP) in urine samples from celiac patients on a gluten-free diet clinically responsive and non-responsive to dietary treatment and from suspected celiac patients already on a gluten-free diet.

DETAILED DESCRIPTION:
Once a year, celiac patients perform a clinical (gastroenterological visit) and blood chemistry (blood tests) check. At the Center for the Prevention and Diagnosis of Celiac Disease, about 1400 check-ups of celiac patients are carried out per year. During this annual control visit, consecutive patients afferent to the center and suffering from celiac disease who have been treated for more than 6 months, clinically "responsive" and "non-responsive" to the gluten free diet (GFD), will be invited to participate in the proposed study. Those who participate will be given the symptom questionnaires (VAS), the food questionnaire in order to evaluate the relevance of the symptoms reported and the type of diet followed by the patient and the adherence test to the gluten-free diet (CDAT). Urine samples will be collected to test the presence of GIP (gluten immunogenic peptides) and for patients whose samples test positive, will be asked for a stool sample to detect GIP.

Subjects with suspected celiac disease but already on a gluten-free diet will undergo a challenge, or the reintroduction of gluten in incremental steps of three weeks (routinely performed as per the instructions of the Italian Health Care System).

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 65 years old
* Gender: Males and Females
* Patients: suffering from Celiac Disease and suspected, but already on a gluten-free diet

Exclusion Criteria:

* Celiac patients less than 6 months after diagnosis
* Celiac patients reporting intentional gluten ingestion

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be patients with celiac disease and suspected celiac disease (about 300)
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2022-02-01 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
GIP | 3 weeks
  GIP Immunogenic Peptide Assay in Urine

SECONDARY OUTCOMES:
Gluten-free diet | 3 weeks
  Assessment of adherence to gluten-free diet and of gluten food intake

CONTACTS AND LOCATIONS:
Overall Officials: Luca Elli, PhD, Principal Investigator — Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico di Milano
Locations (1):
- Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico di Milano, Milan, MI, Italy

REFERENCES:
- [Result] Comino I, Real A, Vivas S, Siglez MA, Caminero A, Nistal E, Casqueiro J, Rodriguez-Herrera A, Cebolla A, Sousa C. Monitoring of gluten-free diet compliance in celiac patients by assessment of gliadin 33-mer equivalent epitopes in feces. Am J Clin Nutr. 2012 Mar;95(3):670-7. doi: 10.3945/ajcn.111.026708. Epub 2012 Jan 18. PMID 22258271
- [Result] Comino I, Fernandez-Banares F, Esteve M, Ortigosa L, Castillejo G, Fambuena B, Ribes-Koninckx C, Sierra C, Rodriguez-Herrera A, Salazar JC, Caunedo A, Marugan-Miguelsanz JM, Garrote JA, Vivas S, Lo Iacono O, Nunez A, Vaquero L, Vegas AM, Crespo L, Fernandez-Salazar L, Arranz E, Jimenez-Garcia VA, Antonio Montes-Cano M, Espin B, Galera A, Valverde J, Giron FJ, Bolonio M, Millan A, Cerezo FM, Guajardo C, Alberto JR, Rosinach M, Segura V, Leon F, Marinich J, Munoz-Suano A, Romero-Gomez M, Cebolla A, Sousa C. Fecal Gluten Peptides Reveal Limitations of Serological Tests and Food Questionnaires for Monitoring Gluten-Free Diet in Celiac Disease Patients. Am J Gastroenterol. 2016 Oct;111(10):1456-1465. doi: 10.1038/ajg.2016.439. Epub 2016 Sep 20. PMID 27644734
- [Result] Moreno ML, Cebolla A, Munoz-Suano A, Carrillo-Carrion C, Comino I, Pizarro A, Leon F, Rodriguez-Herrera A, Sousa C. Detection of gluten immunogenic peptides in the urine of patients with coeliac disease reveals transgressions in the gluten-free diet and incomplete mucosal healing. Gut. 2017 Feb;66(2):250-257. doi: 10.1136/gutjnl-2015-310148. Epub 2015 Nov 25. PMID 26608460